CLINICAL TRIAL: NCT03667378
Title: Evaluating the Impact of Proactive Palliative Care in Patients Initiating Phase I Targeted or Immune-Based Cancer Therapeutics: A Randomized Controlled Trial
Brief Title: Investigating the Impact of Proactive Palliative Care
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-363
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Solid Tumor Cancers; Locally Advanced Solid Tumor Cancers
Keywords: Quality of Life; Supportive Care; 18-363
MeSH Terms: interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- supportive care visits: A concurrent supportive care intervention (intervention arm) Study assessments will be conducted at baseline (t0); at 3-6 weeks +/- 1 week from Day 1 of receiving investigational therapy, prior to sharing information on treatment response and before the first planned scan to evaluate extent of disease (t1); and at 8-12 weeks (the end of the 3 month total study time period) (t2).intervention arm will have at least monthly visits with a supportive care clinician
  Interventions: Behavioral: Expectations Survey (CanCORS); Behavioral: Values Survey (Serious Illness Care Program); Behavioral: Functional Assessment of Cancer Therapy-General (FACT-G); Behavioral: NCCN Distress Thermometer; Behavioral: Hospital Anxiety and Depression Scale (HADS); Behavioral: Quality of Communication (QOC); Behavioral: visits with a supportive care clinician
- without supportive care visits: A concurrent supportive care intervention (intervention arm) Study assessments will be conducted at baseline (t0); at 3-6 weeks +/- 1 week from Day 1 of receiving investigational therapy, prior to sharing information on treatment response and before the first planned scan to evaluate extent of disease (t1); and at 8-12 weeks (the end of the 3 month total study time period) (t2).intervention arm will have at least monthly visits with a supportive care clinicianTo receive the investigational cancer treatment alone (control arm) no monthly visit with a supportive care clinician.
  Interventions: Behavioral: Expectations Survey (CanCORS); Behavioral: Values Survey (Serious Illness Care Program); Behavioral: Functional Assessment of Cancer Therapy-General (FACT-G); Behavioral: NCCN Distress Thermometer; Behavioral: Hospital Anxiety and Depression Scale (HADS); Behavioral: Quality of Communication (QOC)

INTERVENTIONS:
Behavioral: Expectations Survey (CanCORS) — Study assessments will be conducted at baseline (t0); at 3-6 weeks +/- 1 week from Day 1 of receiving investigational therapy, prior to sharing information on treatment response and before the first planned scan to evaluate extent of disease (t1); and at 8-12 weeks (the end of the 3 month total study time period) (t2).
Behavioral: Values Survey (Serious Illness Care Program) — Study assessments will be conducted at baseline (t0); at 3-6 weeks +/- 1 week from Day 1 of receiving investigational therapy, prior to sharing information on treatment response and before the first planned scan to evaluate extent of disease (t1); and at 8-12 weeks (the end of the 3 month total study time period) (t2).
Behavioral: Functional Assessment of Cancer Therapy-General (FACT-G) — Study assessments will be conducted at baseline (t0); at 3-6 weeks +/- 1 week from Day 1 of receiving investigational therapy, prior to sharing information on treatment response and before the first planned scan to evaluate extent of disease (t1); and at 8-12 weeks (the end of the 3 month total study time period) (t2).
Behavioral: NCCN Distress Thermometer — Study assessments will be conducted at baseline (t0); at 3-6 weeks +/- 1 week from Day 1 of receiving investigational therapy, prior to sharing information on treatment response and before the first planned scan to evaluate extent of disease (t1); and at 8-12 weeks (the end of the 3 month total study time period) (t2).
Behavioral: Hospital Anxiety and Depression Scale (HADS) — Study assessments will be conducted at baseline (t0); at 3-6 weeks +/- 1 week from Day 1 of receiving investigational therapy, prior to sharing information on treatment response and before the first planned scan to evaluate extent of disease (t1); and at 8-12 weeks (the end of the 3 month total study time period) (t2).
Behavioral: Quality of Communication (QOC) — Study assessments will be conducted at baseline (t0); at 3-6 weeks +/- 1 week from Day 1 of receiving investigational therapy, prior to sharing information on treatment response and before the first planned scan to evaluate extent of disease (t1); and at 8-12 weeks (the end of the 3 month total study time period) (t2).
Behavioral: visits with a supportive care clinician — Monthly visits with a supportive care clinician
  Groups: supportive care visits

SUMMARY:
This study will test whether adding personalized supportive care to medical treatment on a clinical trial affects the study participants' ability and desire to discuss their symptoms, their concerns about the future, and their approach to coping with cancer. The effects of supportive care on participants' responses to questions about these topics will be compared with those of other study participants who are being treated for cancer in a clinical trial, but are not receiving personalized supportive care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with disease progression on at least one standard chemotherapy regimen, and now eligible and consented to begin Phase I, Phase I/Ib, Phase I/II and non-randomized Phase II (including basket studies) investigational targeted and immune-based therapeutics in MSK medical oncology, EDD, or ITC clinics
* Able to speak, read, and understand English well enough to complete study assessments in the judgment of the consenting professional
* 18 years of age and older
* Has a progressive or metastatic solid tumor cancer with MSK pathology confirmation at the primary or metastatic anatomic site

Exclusion Criteria:

* Patients who already are receiving specialty supportive care (already referred for a supportive care consultation) prior to enrollment in a Phase I protocol.
* Patients will be excluded if the Phase I, Phase I/Ib, Phase I/II or Phase II trial involves known active drugs in combination with experimental drugs, in which the patient has not previously received the known active drug or active drugs of the same class. For example, a patient with metastatic pancreatic cancer who has not received gemcitabine/nab-paclitaxel, but enrolls on a study that tests an experimental drug in addition to gemcitabine/nab-paclitaxel, will be excluded.
* Significant psychiatric or cognitive disturbance in the primary clinician"s or investigator"s judgment, to preclude providing informed consent or participating in the interventions (i.e. acute psychiatric symptoms which require individual treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients with metastatic or locally advanced solid tumor cancers who progress beyond standard treatment and are deemed eligible to receive treatment with investigational targeted or immune-based therapeutics with Phase I, Phase I/Ib, and Phase I/II trials at MSK.
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
patients' expectations for therapeutic benefit | 3 months
  using the CanCORS Expectations Survey, which will assess, on a 4-point Likert-type scale, patients' expectations for therapeutic benefit after talking with their doctors about their experimental drug

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Epstein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm